CLINICAL TRIAL: NCT00777829
Title: Understanding Memory Consolidation by Studying Pharmacologically Enhanced Naps.
Brief Title: Memory Consolidation in Pharmacologically Enhanced Naps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sara C. Mednick, Prinicipal Investigator, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: K01MH080992-01 (NIH); K01MH080992-01 (NIH); 071529; DNBBS 7K-TGNB; NCT00773032 (obsolete NCT alias)
Record Dates: First submitted 2008-10-20; First posted 2008-10-22 (Estimated); Results first posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Sleep
Keywords: Nap; Pharmacology; Memory; Visual Learning; Verbal Memory; Motor Learning
MeSH Terms: conditions — Spatial Learning | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- zolpidem first, then placebo (Experimental): Participants received one dose of zolpidem for one nap, then had a one week washout period, followed by once dose of placebo for one nap.
  Interventions: Drug: zolpidem; Drug: Placebo
- Placebo first, then zolpidem (Placebo Comparator): Participants received one dose of placebo for one nap, then had a one week washout period, followed by once dose of zolpidem for one nap.
  Interventions: Drug: zolpidem; Drug: Placebo

INTERVENTIONS:
Drug: zolpidem — Participants will receive one dose of 10 mg before each nap.
Drug: Placebo — Participants will receive a dose of placebo before each nap.

SUMMARY:
This study will examine whether various drugs affecting sleep cycles can improve different kinds of memory.

DETAILED DESCRIPTION:
Research provides evidence for strong, specific connections between sleeping and memory. This research shows that sleeping is necessary for certain types of memories to form, certain sleep stages lead to specific types of learning and memory consolidation, and naps are as effective as night-time sleep in these learning and memory processes. Current evidence also indicates that there are different types of memory and that the different types can operate and develop independently. In this study, three different memory types will be examined: perceptual, motor, and declarative memory. Perceptual memory is measured through the ability to recognize discrete stimuli; motor memory is measured through the ability to perform specific, coordinated tasks; and declarative memory is measured through the ability to recite memorized information. Different stages in the sleep cycle correlate with improvements in each of these memory processes. For instance, improvement of perceptual memory tasks is dependent on rapid eye motion (REM) sleep; motor learning is related to sleep stage 2; and declarative memory consolidation is related to short wave sleep (SWS), which includes sleep stages 3 and 4.

New drugs can target specific sleep stages and increase the amount of time people spend in those stages when they sleep. For example, the new prescription drug zolpidem increases time spent in stage 2 during sleep, and the drug sodium oxybate increases time spent in SWS. Compared to sleep impacted by either zolpidem or sodium oxybate, normal sleep has proportionally more time spent in REM. This study will use medications, or their lack, to manipulate how much time is spent in REM, stage 2, and SWS. The study will then examine whether the percentage of sleep spent in different stages affects the learning processes associated with those stages.

Participation in this study will last 6 weeks. At the outset, participants will undergo a 2-hour screening visit that will include a medical history, a physical examination, routine lab tests, urine tests for drugs and pregnancy, an electrocardiogram, and a clinical interview for mental health. Participants will also be asked to complete a series of questionnaires on subjective sleep quality, sleep quantity, and daytime sleepiness.

Participants will complete five study visits, beginning 1 week from screening and separated by 5 to 10 days to allow drug wash-out and recovery from effects of the previous visit. Each study visit will involve an overnight stay in a sleep lab. Participants will arrive at 8 PM, go to bed at 10 PM, and be awakened at 5 AM. Between 6 and 8 AM, they will undergo three different tests, each corresponding to a different type of learning and memory process: perceptual, motor, or declarative. The test will include recognizing a target image, typing a specific finger sequence on a keyboard, and verbally recalling a list of words. Participants will receive one of the study drugs or placebo at 8:30 AM and then be allowed to take a 90-minute nap between 9 and 11 AM. They will receive a different drug, different dosage, or placebo at each study visit. Between 4 and 6 PM, they will be retested on the previous three tests. While sleeping, participants will be outfitted with sensors monitoring muscle activity, eye movements, brain waves, heart and lung functioning, and-on the first night-breathing.

For the entire duration of the study, participants will wear an actigraph, which is a wristwatch-like device that monitors sleep cycles. Participants will also be required to maintain a regular sleep schedule, going to sleep and waking up in the same 2-hour window each day. They will also report on sleep schedule and caffeine, alcohol, and drug use in a daily sleep diary. Caffeine, alcohol, and drug use will be prohibited starting at noon on the day prior to each study visit.

ELIGIBILITY:
Inclusion Criteria:

* Speaks English
* Resides in the general San Diego community
* Completed at least 12 years of formal education, because education may affect performance on the cognitive task

Exclusion Criteria:

* No regular sleep-wake schedule, defined as not meeting study criteria or scoring between 31 and 69 on the Horne-Ostberg Morningness-Eveningness Questionnaire
* Presence of a sleep disorder reported or detected on the questionnaires
* Personal or immediate family (i.e., first degree relative) history of diagnosed significant psychopathology
* Personal history of head injury with loss of consciousness for more than 15 minutes or with seizures
* History of substance dependence
* Current use of any psychotropic medications
* Any cardiac, respiratory, or other medical condition that may affect cerebral metabolism
* Noncorrectable vision and audition impairments

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-09-01 (Actual); Primary Completion 2011-06-01 (Actual); Study Completion 2011-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara C. Mednick, PhD, Principal Investigator — UCSD
Locations (1):
- UCSD General Clinical Research Center Laboratory for Sleep and Chronobiology (GCRC-LSC), La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zolpidem First, Then Placebo | Placebo First, Then Zolpidem
Started | 15 | 15
Study Orientation | 15 | 13
Completed | 15 | 13
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Participants: This was a within-subjects design, so all 30 started in the participant flow, but only 28 completed all arms of the study.
Arm/Group | All Participants
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Pharmacological Enhancement of Specific Sleep Parameters
Description: Number of sleep spindles comparing placebo vs active drug. We count spindles in the EEG record.
Time Frame: Two weeks
Measure: Mean (Standard Deviation); unit: sleep spindles
Groups:
- Zolpidem: This arm reflects all participants who received the drug (one dose of 10mg before each nap) during the entire course of the study.
- Placebo: This arm reflects all participants who received the placebo (a dose of placebo before each nap) during the entire course of the study.
Arm/Group | Zolpidem | Placebo
Number analyzed (Participants) | 28 | 28
sleep spindles | 3 (0.5) | 1 (0.5)

2. Secondary Outcome: Correlation of Pharmacological Interventions With Sleep-stage-specific Memory Tasks
Description: improvement on a verbal memory task in active drug. We measured the number of words recalled.
Time Frame: two weeks
Measure: Mean (Standard Deviation); unit: recall of words
Groups:
- Zolpidem: This arm reflects all participants who received the drug (1 dose of 10mg before each nap) during the entire course of the study.
- Placebo: This arm reflects all participants who received the placebo (1 dose of placebo before each nap) during the entire course of the study.
Arm/Group | Zolpidem | Placebo
Number analyzed (Participants) | 28 | 28
recall of words | 3 (1.0) | 1 (0.5)

ADVERSE EVENTS:
Arm/Group | Zolpidem | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 17/28 | 0/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zolpidem (N=28) | Placebo (N=28)
drowsiness (General disorders) | 17 | 0
dizziness (General disorders) | 12 | 0
nausea (General disorders) | 4 | 0
vomiting (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No